CLINICAL TRIAL: NCT00969488
Title: The Effect of a High Protein Diet on Body Weight Change and Body Composition During Post-partum: Randomized Clinical Trial Study
Brief Title: The Effect of a High Protein Diet on Body Weight Change During Post-partum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Rosely Sichieri, Universidade do Estado do Rio de Janeiro. Departamento de Epidemiologia
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Pensa Rio - UERJ/FAPERJ
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2009-08

CONDITIONS: Overweight
Keywords: matern diet; obese; postpartum; body weight change; Women with overweight
MeSH Terms: conditions — Overweight; Obesity; Body Weight Changes | interventions — Diet, High-Protein

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high protein diet group (Experimental): Women in high protein diet will be stimulate to consumption of high protein foods and restrict the consumption of carbohydrates in the experimental group. The women in the intervention group will be incentivized to substitute breads and pastas for high protein foods (legumes, milk and its derivatives, eggs, fish, and lean meats). The experimental groups will also receive six cans of sardine to increase the women's commitment to the study.
  Both women group will receive a nutritional plan based on an 1800 kcal diet.
  Interventions: Other: High protein diet
- normal protein diet group (Active Comparator): The control group will receive a diet to lose weight with norma protein intake and will receive 2kg of pasta to increase the women's commitment to the study. The nutritional plan based on an 1800 kcal diet.
  Interventions: Other: High protein diet

INTERVENTIONS:
Other: High protein diet — INTERVENTION is to stimulate the consumption of high protein foods and restrict the consumption of carbohydrates in the experimental group.
  The women in the intervention group will be incentivized to substitute breads and pastas for high protein foods (legumes, milk and its derivatives, eggs, fish, and lean meats).
  Other Names: High protein diet group; Normal protein diet group

SUMMARY:
Nearly 20% of women do not return to their pré-gestacional body weight. The purpose of this study is to investigate the effect of diet and socio-demographics factors during gestation and postpartum period to body weight change after delivery. This is a clinical trial with 180 women interviewed at 1 (baseline), 2, 3, 4, 5 and 6 months postpartum. The dietary data were obtained by employing the Food Consumption Frequency Questionnaire with reference to the first and sixth months of postpartum.

DETAILED DESCRIPTION:
SUBJECTS AND METHODS

1. STUDY DESIGN AND SUBJECTS This randomized clinical trial study examined the efficacy of two weight loss diets with different intake of protein by kg of body weight in postpartum women that had at Hospital Leonel de Moura Brizola do Município de Mesquita, situated at Rio de Janeiro State. Inclusion criterion were women with body mass index (BMI) ≥ 26 kg/m2, age between 18 and 45 years, without chronic illnesses (thyroid disease).
2. COLLECTION OF DATA:

2.1- Collection: Maternity. The women with BMI ≥ 26 kg/m2 are invited to participate in the study at the maternity until 3 days after child birth. The women that chose to participate will be scheduled to come in for their first visit approximately one month after the birth of their child. The visits will occur in the Hospital Municipal Leonel de Moura Brizola and the evaluations of body composition by DXA will take place at the University of the Rio de Janeiro State. The room at the University prepared for the visits will provide comfort for the mothers and their babies. The place picked for the participants of this study is the hospital at which the sponsor works and because it consists of low income women with high risk of obesity post partum.

In this occasion, dietary intake, antropometrics and socio-demographic measures were been taken. The women will answer their clinical history, foodnutrient intake of the last six months prior to the birth of their child, breastfeeding, their social-demographics status, and life style (education, civil state, age, work, living conditions, race, smoking, and consumption of alcohol). The participant's race will be determined by skin color given by the participants themselves as well as the interviewer. Body weight and composition and height will be measured using an electronic scale (Tanita, Model BWB-627A) stadiometer (Holtain Limited, Crymych, United Kingdom), respectively.

2.2- First month of postpartum: cohort baseline. At this moment, the women will receive information about the study, the procedures that will take place, the objectives of the study, and will sign the terms of consent. Only the women that show up to this visit will form the cohort for the randomized diet. The participants of the study will be allocated randomly into a control and experimental group. After the allocation, the women will receive a program to lose weight as will be discussed in section 3- Intervention.

The body weight and body composition of the participants will be measured on the first interview and all others waves of follow-up with an electronic scale (Tanita, Model BWB-627A) that has a capacity 150kg and precision of 0.1kg.

All of the participants will receive nutritional guidance. The mothers will be guied to the Mesquita's reference laboratorie to collect blood samples and diagnose any nutritional deficiencies or physiological alterations of the reproductive period.

The dietary intake will be obtained by a 24-hour recall and a semiquantitave food frequency questionnaire (FFQ) previously validated by Sichieri e Everhart (1998), about the last month diet. The is used in epidemiological studies and more specifically to evaluate post partum mothers (Rodrigues & Costa, 2001, Kesa & Oldewagw-Theron, 2004, George et al., 2005). Studies have shown that this instrument is valid and reproducible to measure nutrients intake (Erkkola et al., 2001; Bunin et al., 2001). Questions about physical activity, breastfeeding and perception of body composition will be done in this visit. The evaluation of physical activity will be obtained through a questionnaire of leisure physical activities that has been previously validated (Pardini et al., 2000). At this visit, the women will indicate in a scale of body perception, which women model they perceive to be closest to their own body.

2.3-Second Month post partum: second wave of follow-up. The women will be transported to UERJ for their second visit. At this visit, the women's weight, body perimeters, and skin folds. Body composition will be determined through bioimpedância (Biodynamics 450) and by the DXA which scans the entire body transversely in sections of low and high energy X rays of 1cm. At each section of the body that is scanned, the body's composition of body fat and lean mass will be determined. This method has been termed as the most accurate and precise device for measuring body composition (Lohman & Chen, 2005). The DXA will quantify the lean mass, bone mass, body fat, and abdominal fat. The total body fat will be expressed in terms relative to body mass. The use of the DXA is conditioned to a negative pregnancy test.

The DXA is an accurate non invasive method of low radiation (1/10 do Raio-X) (Ellis et al., 1994; Tataranni & Ravussin, 1995; Marques et al., 2000) that is widely used to evaluate the density of bone minerals in adults (Paton et al., 2003), newborns (Jarjou et al., 2006), lactating women (Richie et al, 1998; Laskey et al., 1998; Bezerra et al., 2004), and also in the evaluation of body composition and percentage of body fat (Kim et al., 2002; Rech et al., 2006).

In this visit the women will answer breastfeeding, social and diet commitment questionnaires.

2.4-Third month postpartum: third wave of follow-up. The participants will once again be weighted and answer a 24-hour recall. Information about the mother's breast-feeding and commitment to the diet will be obtained. A questionnaire tracking the mother's commitment to the diet has been formulated based on the analysis of the variation of the diet quality of the pregnant women. (Castro et al., 2006; Castro et al., no prelo). The nutrients responsible for the difference in the density of the diet are: rice, beans, vegetables, fruits, cereals, meats, poultry, milk, milk derivatives, sweets, coffee, wine, and beer. Since the study is based on overweight women and in which the intervention is based on a high protein diet: sardines, fish, eggs, sodas, and finger foods were inserted into the questionnaire. Some food items grouped into cereals were placed separately on the questionnaire in order to analyze the differences of carbohydrate consumption in the groups of: pasta, breads, cookies, cakes, potatoes, yucca, and yams.

At this visit, the women will respond to a psychological questionnaire that will be used to evaluate minor psychiatric disturbance prior to the reproductive cycle and the Edimburgo scale to evaluate postpartum depression. The women will once again evaluate themselves on the body perception scale and will be guied to collect the second blood sample.

2.5-Fourth month postpartum: fourth wave of follow-up. In the fourth month's visit, the participants will be evaluated on their weight, body perimeters and the measurements of body composition, breastfeeding and questionnaire of diet commitment. The 24- hour recall diet will be obtained.

2-6- Fifth month postpartum: fifth wave of follow-up. The weight of the mothers and their babies will be taken as well as an evaluation of their body's composition based on bioimpedância measurements and body perimeters. Information of breast-feeding will be collected along with another 24-hour food intake recall, FFQ, physical activity, and the body perception scale. A final blood sample will be collected and compared with the initial nutritional state. Information about the women's commitment to the diet and depression will also be obtained.

2-6- Sixth month postpartum: sixth wave of follow-up. The women will be transported to UERJ for their sixth visit. The mother and child's weight will be evaluated in this occasion. Body composition will be taken by dual-energy X-ray absorptiometry (DXA). Antropometrics measuraments (circumferences and skin folds) will be obtained as recommended by Lohman (1988). In this visit the women will be evaluated on their waist and hip circumferences measured by World Health Organization (1997) and will answer breastfeeding, social and diet commitment questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women with body mass index (BMI) ≥ 26 kg/m2
* Age between 18 and 45 years

Exclusion Criteria:

* Chronic illnesses (thyroid disease)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Body weight change | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosely Sichieri, Phd, Principal Investigator — Rio de Janeiro State University; Maria B Castro, Phd, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Hospital Municipal Leonel de Moura Brizola, Mesquita, Rio de Janeiro, Brazil